CLINICAL TRIAL: NCT02000947
Title: A Phase 1b Open-label Study to Evaluate the Safety and Tolerability of MEDI4736 in Combination With Tremelimumab in Subjects With Advanced Non-small Cell Lung Cancer
Brief Title: A Phase 1b Study of MEDI4736 in Combination With Tremelimumab in Subjects With Advanced Non-small Cell Lung Cancer
Acronym: D4190C00006
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4190C00006; 2015-003715-38 (EudraCT Number)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: NSCLC; Non-small Cell Lung Cancer; Lung Cancer
Keywords: anti-CTLA-4; anti-PD-L1; immunotherapy; IMTC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): MEDI4736 and tremelimumab received by intravenous infusion.
  Interventions: Drug: MEDI4736; Drug: Tremelimumab
- Arm A (Experimental): Medi4736 and tremelimumab received by intravenous infusion
  Interventions: Drug: MEDI4736; Drug: Tremelimumab
- Arm B (Experimental): MEDI4736 and tremelimumab received by intravenous infusion
  Interventions: Drug: MEDI4736; Drug: tremelimumab
- Arm C (Experimental): MEDI4736 and tremelimumab received by intravenous infursion
  Interventions: Drug: MEDI4736; Drug: tremelimumab

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 is an anti-PD-L1 monoclonal antibody (MAb).
Drug: Tremelimumab — Tremelimumab is an anti-CTLA4 monoclonal antibody (mAb).
  Arms: Arm A; Dose Escalation
Drug: tremelimumab — Tremelimumab is an anti-CTLA4 monoclonal antibody (mAb).
  Arms: Arm B; Arm C

SUMMARY:
The purpose of this study is to determine if MEDI4736 will be adequately tolerated in combination with tremelimumab in subjects with advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation, and dose expansion study of MEDI4736 in combination with tremelimumab to evaluate the safety, tolerability, pharmacokinetic (PK), immunogenicity, and antitumor activity of MEDI4736 in combination with tremelimumab in adult subjects with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Advanced non-small cell lung cancer
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
4. Adequate organ and marrow function

Exclusion Criteria:

1. Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment
2. Current or prior use of immunosuppressive medication within 14 days before the first dose of study drugs
3. Active or prior documented autoimmune disease within the last 2 years.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting adverse events | Screening through 90 days after the last dose of study medication
  The number of subjects reporting adverse events (AEs) and number (percentage) of subjects reporting serious adverse events (SAEs) as graded by CTCAE Version 4.03
Objective response | At least 24 weeks as compared to baseline
  Best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as defined as the best response among all overall responses recorded from the start of treatment until progression, or the last evaluable disease assessment in the absence of progressive disease (PD) prior to the initiation of subsequent anti-cancer therapy, or discontinuation from the study, whichever occurs first.
Number of subjects experiencing dose-limiting toxicities (DLTs) | Depending upon the cohort, the DLT evaluation period is from the 1st dose of study medication until (1) the 3rd dose of MEDI4736 and tremelimumab (2) the 2nd dose of MEDI4736 and tremelimumab or (3) the 3rd dose of MEDI4736 and 2nd dose of tremelimumab
  The maximum tolerated dose (MTD), which is the highest dose within a cohort where no more than 1 out of 6 subjects experience DLTs or the highest protocol-defined dose for each agent in the absence of exceeding the MTD, will be evaluated using the following safety assessments: adverse events, serious advents, laboratory evaluations, vital signs, physical examinations, and electrocardiogram (ECG) results. Measurements will be aggregated to determine whether a subject has experienced a DLT as assessed by the investigator.

SECONDARY OUTCOMES:
Immunogenicity of tremelimumab in combination with MEDI4736 | During treatment through study completion, about 2 years
  Immunogenicity of MEDI4736 and tremelimumab will include the number and percentage of subjects who develop detectable anti-drug antibodies (ADAs).
Antitumor activity of tremelimumab in combination with MEDI4736 | During treatment through study completion, about 2 years
  Antitumor activity will include objective response (OR) and disease control (DC) based on RECIST Version 1.1, duration of response (DoR), progression-free survival (PFS), and overall survival (OS).
Pharmacokinetic parameters | During treatment through study completion, about 2 years
  Assessment of PK of MEDI4736 and tremelimumab will include individual MEDI4736 and tremelimumab concentrations in serum, and PK parameters including peak concentration (Cmax), area under the concentration-time curve (AUC), clearance (CL), and half-life (t½).
Number of subjects reporting adverse events | Screening through 90 days after the last dose of study medication
  The number of subjects reporting adverse events (AEs) and number (percentage) of subjects reporting serious adverse events (SAEs) as graded by CTCAE Version 4.03

OTHER OUTCOMES:
Biomarkers | During treatment through study completion, about 2 years
  To evaluate biomarkers that may correlate with clinical activity of MEDI4736 in combination with tremelimumab

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (59):
- United States (25):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Tampa, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Lebanon, New Hampshire
  - Research Site, New York, New York
  - Research Site, Huntersville, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
- Australia (3):
  - Research Site, Darlinghurst
  - Research Site, Gosford
  - Research Site, Kogarah
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Liège
- France (8):
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, La Tronche
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Saint-Herblain
- Italy (6):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Rozzano
  - Research Site, Saronno
  - Research Site, Siena
  - Research Site, Sondrio
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Jaén
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Derived] Garon EB, Spira AI, Goldberg SB, Chaft JE, Papadimitrakopoulou V, Cascone T, Antonia SJ, Brahmer JR, Camidge DR, Powderly JD, Wozniak AJ, Felip E, Wu S, Ascierto ML, Elgeioushi N, Awad MM. Brief Report: Safety and Antitumor Activity of Durvalumab Plus Tremelimumab in Programmed Cell Death-(Ligand)1-Monotherapy Pretreated, Advanced NSCLC: Results From a Phase 1b Clinical Trial. J Thorac Oncol. 2023 Aug;18(8):1094-1102. doi: 10.1016/j.jtho.2023.04.020. Epub 2023 May 4. PMID 37146752
- [Derived] Antonia S, Goldberg SB, Balmanoukian A, Chaft JE, Sanborn RE, Gupta A, Narwal R, Steele K, Gu Y, Karakunnel JJ, Rizvi NA. Safety and antitumour activity of durvalumab plus tremelimumab in non-small cell lung cancer: a multicentre, phase 1b study. Lancet Oncol. 2016 Mar;17(3):299-308. doi: 10.1016/S1470-2045(15)00544-6. Epub 2016 Feb 6. PMID 26858122